CLINICAL TRIAL: NCT04572490
Title: The Comparison of Narrow and Regular Platform Dental Implants Placed Posterior Regions
Brief Title: Comparison of Narrow and Regular Implants
Status: Completed | Type: Observational
Sponsor: T.C. Dumlupınar Üniversitesi (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assist Prof, T.C. Dumlupınar Üniversitesi
Other Study IDs: 2019/07-4
Record Dates: First submitted 2020-09-24; First posted 2020-10-01 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Dental Implant Failed; Alveolar Bone Loss; Complication,Postoperative
Keywords: Dental implants Alveolar bone loss
MeSH Terms: conditions — Alveolar Bone Loss; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Narrow platform implant: All measurements will be obtained after dental implant functional loading. Periodontal index will be recorded and alveolar bone loss measurements will be made on periapical radiographs.
  Interventions: Diagnostic Test: periapical radiograph
- Regular platform implants: All measurements will be obtained after dental implant functional loading. Periodontal index will be recorded and alveolar bone loss measurements will be made on periapical radiographs.
  Interventions: Diagnostic Test: periapical radiograph

INTERVENTIONS:
Diagnostic Test: periapical radiograph — alveolar bone loss measurement on standardized parallel periapical radiograph

SUMMARY:
The study was designed as a retrospective, parallel, two years longitudinal pilot trial. Twenty-eight patients (mean age: 48.34 ± 6.06) aged between 35 and 60 years and 66 TiUnite surfaces (Nobel Biocare Parallel Conical Connection), bone level dental implant were included in the study. The implants were divided into two different groups according to the NPIs and regular platform implants(RPIs). The mean implant lengths, plaque index(PI), gingival index(GI), periodontal pocket depth(PD), gingival recession(GR), keratinized gingival width(KGW) and bleeding on probing(BOP) values were recorded. The Student's t-test used for between-group comparison.

DETAILED DESCRIPTION:
Fifty-one participants and 123 dental implants were evaluated; twenty-three participants and 49 dental implants were excluded because of the different commercial brand dental implant (AstraTech, Straumann Roxolid, Bilimplant) and declining to participate. Seventy-four TiUnite dental implants were included in the study, but 8 TiUnite surface implants placed in the anterior region were excluded. Consequently, 15 male and 13 female patients and 66 dental implants were included in the study. This randomized retrospective clinical trial was designed according to the Consolidated Standards of Reporting Trials (CONSORT) Statement guidelines. A CONSORT Flow Chart of this study was shown in Figure 118.

The assignment was performed according to the dental implant diameters to include cases in the NPI and RPI which are the test and control groups. All dental implants involved are the Nobel Biocare Parallel CC brand (Nobel Biocare, Gothenburg, Sweden) with a TiUnite surface, and it defined a regular diameter of 4.3 mm and narrow diameter of 3.75 mm. Dental implants divided into two groups according to implant diameter, the NPI group comprised 3.75 mm diameter (NP, Ø= 3.75 mm) implants, and the RPI group comprised 4.3 mm diameter (RP, Ø= 4.3mm) implants (implant lengths: 10 mm-13 mm).

Clinical Measurements The clinical measurements were recorded at follow-up sessions using a periodontal probe that was calibrated in 1 mm increments. The clinical measurements were as follows: 1) plaque index (PI); 2) gingival index (GI); 3) probing depth (PD), the distance between the gingival margin and the bottom of a pocket; 4) clinical attachment level (CAL); the distance from the neck of the implant and the bottom of the pocket; 5) bleeding on probing (BOP); 6) keratinized gingival width (KGW), the height of peri-implant keratinized mucosa; 7) gingival recession (GR), the distance between the neck of the implant and the gingival margin. The same researcher performed all clinical measurements. A calibration protocol was applied to the reliability of measurements. PI, GI, PD, CAL, GR, KGW meaurements on five patients and ten peri-implant values were assessed. Calibration was accepted when measurements were 90% similar20. All clinical measurements were recorded for four sites (mesiobuccal, distobuccal, mid-buccal, mesiopalatal, midpalatal, and distopalatal) per peri-implant region. PD and PI measurements are reliable in peri-implantitis diagnosis21.

Prosthetic complications of patients were also evaluated clinically. Veneer ceramic chipping, abutment screw loosening or fracture, implant fracture, loss of retention were recorded.

Radiographic Measurements The studies have reported that periapical radiographs taken with the parallel technique are reliable in determining the MBL changes at different follow-ups. Digital periapical radiographs of the posterior region were obtained using a parallel method at follow-up sessions. MBL measurements were provided on periapical radiographs by a software program (Mediadent Software, The Dental Imaging Company, London, England). Ten radiographic MBL measurements around peri-implant were performed twice with an interval of 3 weeks, and researcher calibration was accepted when measurements were similar as %90. MBL was measured separately from the mesial and distal parts and also which the average of the two measurements. The reference points for the assessments are the implant shoulder and the most apical end-point of the bone-implant contact point. The vertical length between these two points is defined as MBL.

ELIGIBILITY:
Inclusion Criteria:

* the presence of a dental implant treated with fixed prosthetic restoration placed in the posterior jaw followed for at least one year after functional loading,
* no active periodontal disease,
* no history of penicillin allergy -
* no radiotherapy to the head and neck region
* smoking less than ten cigarettes per day,
* no bone augmentation surgery before or during dental implant surgery,
* aged over 18,
* mesial or distal additional crown restoration was not performed,
* no use of medications that affect bone metabolism and
* not pregnant or lactating.

Exclusion Criteria:

* the implants placed in the anterior region,
* immediate placing and loading
* augmented before or using a graft membrane with surgery

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All dental implants involved are the Nobel Biocare Parallel CC brand (Nobel Biocare, Gothenburg, Sweden) with a TiUnite surface, and it defined a regular diameter of 4.3 mm and narrow diameter of 3.75 mm. Dental implants divided into two groups according to implant diameter, the NPI group comprised 3.75 mm diameter (NP, Ø= 3.75 mm) implants, and the RPI group comprised 4.3 mm diameter (RP, Ø= 4.3mm) implants (implant lengths: 10 mm-13 mm).
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Marginal bone loss | change from baseline marginal bone loss at postoperatively 24. month
  Peri-implant alveolar bone loss measurements on software program

SECONDARY OUTCOMES:
Keratinized gingival width | change from baseline peri-implant keratinized gingival width at postoperatively 24. month
  Peri-implant keratinized gingival width measurements with clinically

CONTACTS AND LOCATIONS:
Overall Officials: Berceste Guler, PhD, Principal Investigator — Kütahya Health Sciences University
Locations (1):
- Kütahya Health Sciences University Faculty of Dentistry, Kütahya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No